CLINICAL TRIAL: NCT01206582
Title: A Pilot Study of Hemin Therapy for Gastroparesis
Brief Title: A Pilot Study of Hemin Therapy for Gastroparesis (Diabetes Mellitus)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); RECORDATI GROUP (Industry)
Responsible Party: Principal Investigator, Adil Bharucha, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-000129; P01DK068055 (NIH); UL1TR000135 (NIH)
Record Dates: First submitted 2010-09-20; First posted 2010-09-22 (Estimated); Results first posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-01

CONDITIONS: Gastroparesis; Diabetes Mellitus
MeSH Terms: conditions — Gastroparesis; Diabetes Mellitus | interventions — Hemin; Albumins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hemin (Active Comparator): Panhematin®, Ovation Pharmaceuticals, Deerfield, Illinois (IL). Hemin was diluted in 25% albumin to obtain a concentration of 2.4 mg/mL and administered at a dose of 1.25 mL/Kg and at a rate of 60 mL/hour. 10 iv infusions for 8 weeks
  Interventions: Biological: Hemin
- Albumin (Placebo Comparator): 10 iv infusions for 8 weeks
  Interventions: Biological: Albumin

INTERVENTIONS:
Biological: Hemin — 10 iv infusions for 8 weeks
  Other Names: Panhematin®, (Ovation Pharmaceuticals, Deerfield, IL)
  Arms: Hemin
Biological: Albumin — 10 iv infusions for 8 weeks
  Other Names: Albumin (Human) 25% Solution manufactured by CSL Behring.
  Arms: Albumin

SUMMARY:
This study is designed to learn if hemin can increase the production of heme oxygenase 1 and improve gastric (stomach) emptying and symptoms in diabetic patients with slow gastric emptying (gastroparesis).

DETAILED DESCRIPTION:
Therapeutic options for management of diabetic gastroparesis are limited. Failure to maintain upregulation of heme oxygenase 1 (HO1) leads to loss of interstitial cells of Cajal and delayed gastric emptying in diabetic non-obese diabetic mice.

HO1 is an enzyme which protects cells from physical, chemical, and biologic stress. In mice with diabetes and slow gastric emptying, hemin increases HO-1 activity and improves gastric emptying. Hemin is produced from red blood cells and is approved by the Food and Drug Administration for treating acute porphyria, which is an inherited condition caused by an enzyme deficiency. Hemin is not approved by the Food and Drug Administration for treating gastroparesis.

In this study subjects were randomized to intravenous hemin, prepared in albumin, or albumin alone. After infusions on days 1, 3, and 7, weekly infusions were administered for 7 weeks. Assessments included blood tests for HO1 protein and enzyme activity levels, gastric emptying with 13^C-spirulina breath test, autonomic functions (baseline and end), and gastrointestinal symptoms every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

Where relevant (i.e., for ensuring safety), the inclusion and exclusion criteria are similar to those in a recently completed trial of hemin therapy for myelodysplastic syndrome at Rush University, Chicago (http://clinicaltrials.gov/ct2/show/NCT00467610).

* Upper gastrointestinal symptoms which satisfy criteria for postprandial distress syndrome or vomiting for the last 3 months with symptom onset at least 6 months prior to diagnosis
* At least moderately severe symptoms as manifest by a total symptom score of 2.5 or higher on the Gastroparesis Cardinal Symptom Index (GCSI)21
* Delayed gastric emptying (i.e, < 40% emptying at 2 and/or < 90% emptying at 4 hours by scintigraphy)
* No structural cause for symptoms by endoscopy within the past 12 months
* Patient must have a platelet counts > 50,000/microliters and absolute neutrophil counts (ANC) >500/microliters.
* Patient must have adequate hepatic and renal functions, defined as serum bilirubin, serum glutamic-oxaloacetic transaminase (SGOT), and serum glutamate pyruvate transaminase (SGPT) ≤ 2 times the upper limit of normal (ULN), and creatinine ≤ 1.5 times the ULN.
* Able to provide written informed consent before participating in the study

If female:

* Either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or if of childbearing potential, must comply with an effective method of birth control acceptable to the investigator during the study (oral contraceptives, Depo-Provera, intra-uterine device or barrier methods)
* Patient is not breastfeeding.
* Patient of childbearing potential must have a negative urine or serum pregnancy test during the screening period.

Exclusion Criteria:

* History of allergic reaction or significant sensitivity to Panhemantin ®
* Patients who have taken or used any investigational drug or device in the 30 days prior to screening
* Predominant symptoms of epigastric pain or rumination syndrome
* Structural cause for symptoms on recent endoscopy
* Patients with preexisting blood coagulation abnormalities
* Patients with previously documented renal impairment defined as above 150 mmol/L or 1.7 mg/dL serum creatinine
* Previous gastric or intestinal surgery - patients with enteral feeding tubes and/or venting/feeding gastrostomy will be eligible provided they can comply with study requirements. Tube feeding will be stopped 24 hours before the gastric emptying study
* Current use of narcotics, anticholinergic agents (e.g., hyoscyamine, belladonna), anticoagulants (e.g., warfarin) or erythromycin. Gastrointestinal prokinetic drugs (eg metoclopramide, or domperidone) may be continued at a stable dose throughout the study
* History of a pre-existing medical condition that, in the opinion of the investigator, will interfere with the participation in the study.
* History of venous thrombosis or hypercoagulable state
* Poor peripheral venous access, if central venous access is not available
* Uncontrolled active infection
* Any other condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study.
* Known intolerance or allergy to eggs
* Screening weight greater than 130 kg

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adil E Bharucha, MBBS, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at Mayo Clinic in Rochester, Minnesota between Mayo 2010 and November 2013.
Period: Overall Study
Arm/Group | Hemin | Albumin
Started | 11 | 9
Completed | 9 | 7
Not Completed | 2 | 2
Not completed — Withdrew prior to study | 1 | 0
Not completed — Discontinued intervention before week 8 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Hemin: Panhematin®, Ovation Pharmaceuticals, Deerfield, IL. Hemin was diluted in 25% albumin to obtain a concentration of 2.4 mg/mL and administered at a dose of 1.25 mL/Kg and at a rate of 60 mL/hour. 10 iv infusions for 8 weeks
- Total: Total of all reporting groups
Arm/Group | Hemin | Albumin | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (14.4) | 35.2 (14.9) | 41.1 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Venous Plasma Heme-oxygenase 1 (HO1) Protein Concentration
Description: HO1 protein concentration levels in plasma were assessed with a HO1 (human) enzyme-linked immunosorbent assay (ELISA) kit.
Time Frame: baseline, day 3, day 7, day 56
Population: Total number of subjects analyzed varied per time period due to discontinuations, subject and data availability. Subjects analyzed are presented per category as (n=hemin, albumin arms).
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Hemin | Albumin
Number analyzed (Participants) | 11 | 9
ng/mL
  baseline (n=11, 8) | 1.6 (0.3) | 1.5 (0.1)
  Day 3 (n=10, 8) | 10.6 (2.3) | 1.5 (0.3)
  Day 7 (n=8, 8) | 7.0 (2.1) | 1.2 (0.2)
  Day 56 (n=9, 4) | 2.6 (0.8) | 1.0 (0.1)
Statistical Analysis 1: Comparison: Hemin vs Albumin; Comparison for day 3; Test type: Superiority or Other; p = 0.0002, ANCOVA
Statistical Analysis 2: Comparison: Hemin vs Albumin; Comparison for day 7; Test type: Superiority or Other; p = 0.008, ANCOVA

2. Primary Outcome: Venous Monocyte HO1 Activity
Description: HO1 activity in white blood cells was measured by an assay that measures bilirubin production as a marker of HO1 activity.
Time Frame: baseline, Day 3, Day 7, Day 56
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pmol bilirubin/mg/h
Arm/Group | Hemin | Albumin
Number analyzed (Participants) | 11 | 9
pmol bilirubin/mg/h
  Baseline (n=10, 8) | 38.5 (12.0) | 42.1 (10.9)
  Day 3 (n=9, 8) | 373.9 (82.8) | 48.1 (12.9)
  Day 7 (n=8, 8) | 126.2 (51.3) | 36.1 (12.0)
  Day 56 (n=8, 4) | 30.1 (12.7) | 60.1 (23.0)
Statistical Analysis 1: Comparison: Hemin vs Albumin; Comparison for day 3; Test type: Superiority or Other; p = 0.0003, ANCOVA

3. Primary Outcome: Gastric Emptying Half-time
Description: The time for half of the ingested solids or liquids to leave the stomach. Gastric emptying was assessed with ^13C Spirulina Breath Test. After an overnight fast, subjects consumed the test meal containing ^13C Spirulina. Breath samples were collected in duplicate glass tube using a straw to blow into the bottom of the tube to displace contained air. The ^13CO_2 content of the breath was determined by AB Diagnostics. The provide of ^13CO_2 excretion is used to estimate the half-time of gastric emptying.
Time Frame: baseline, day 3, day 7, day 56
Population: as for outcome 1
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Hemin | Albumin
Number analyzed (Participants) | 11 | 9
minutes
  Baseline (n=10, 9) | 161.8 (6.7) | 160.1 (16.3)
  Day 3 (n=10, 9) | 155.6 (9.1) | 155.4 (16.5)
  Day 7 (n=9, 8) | 154.0 (6.5) | 155.4 (15.0)
  Day 56 (n=9, 6) | 161.2 (6.2) | 153.4 (16.4)

4. Secondary Outcome: Gastrointestinal Symptoms
Description: Subjects recorded their GI symptoms every day in the validated Gastroparesis Cardinal Symptom Index (GCSI) - Daily Diary. For each subject, the daily GCSI data were averaged per week. Components coded 0 (no symptoms) to 5 (very severe). GCSI total score is the average of 9 components from the nausea/vomiting, fullness/early satiety, and bloating subscores. These individual subscores are averages of 3,4, and 2 components, respectively. Subscores for upper and lower abdominal pain, heartburn/regurgitation and FDA nausea, vomiting, fullness, and pain (NVFP) composite are averages of 2, 2, 7, and 4 components, respectively.
Time Frame: baseline, 8 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Hemin | Albumin
Number analyzed (Participants) | 9 | 9
units on a scale
  Baseline GCSI total score (n= 9, 9) | 3.1 (0.3) | 3.3 (0.1)
  8 weeks GCSI total score (n=9, 7) | 1.4 (0.3) | 1.9 (0.5)
  Baseline nausea/vomiting subscore (n=9, 9) | 2.9 (0.6) | 3.2 (0.4)
  8 weeks nausea/vomiting subscore (n=9, 7) | 1.3 (0.4) | 1.3 (0.4)
  Baseline fullness/early satiety subscore (n= 9, 9) | 3.8 (0.3) | 3.4 (0.3)
  8 weeks fullness/early satiety subscore (n=9, 7) | 1.9 (0.4) | 2.1 (0.5)
  Baseline bloating subscore (n=9, 9) | 2.6 (0.5) | 3.4 (0.4)
  8 weeks bloating subscore (n=9, 7) | 1.0 (0.3) | 2.4 (0.7)
  Baseline upper abdominal pain score (n= 9, 9) | 3.7 (0.4) | 2.8 (0.6)
  8 weeks upper abdominal pain score (n=9, 7) | 1.4 (0.4) | 1.7 (0.6)
  Baseline lower abdominal pain subscore (n=9, 9) | 2.6 (0.4) | 1.9 (0.4)
  8 weeks lower abdominal pain subscore (n=9, 7) | 1.3 (0.4) | 1.4 (0.5)
  Baseline heartburn/regurgitation subscore (n=9, 9) | 2.0 (0.4) | 1.8 (0.4)
  8 weeks heartburn/regurgitation subscore (n=9, 7) | 1.0 (0.4) | 0.9 (0.5)
  Baseline FDA NVFP composite subscore (n=9, 9) | 3.4 (0.4) | 3.3 (0.2)
  8 weeks FDA NVFP composite subscore (n=9, 7) | 1.5 (0.4) | 1.7 (0.4)

5. Secondary Outcome: Autonomic Functions
Description: Subjects completed a standardized autonomic symptom questionnaire, the Composite Autonomic Severity Score (CASS) which consists of 2 subscores: cardiovagal (CASS-vag; 0-3) and adrenergic (CASS-adr;0-3), where 0, 1, 2, 3 represent non, mild, moderate, and severe dysfunction, respectively.
Time Frame: baseline, Day 56
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Hemin | Albumin
Number analyzed (Participants) | 11 | 9
units on a scale
  CASS vagal score - baseline (n=9, 8) | 1.6 (0.5) | 1.7 (1.1)
  CASS vagal score - day 56 (n=9, 8) | 1.2 (0.4) | 1.9 (0.4)
  Cass adrenergic score - baseline (n=5, 6) | 1.0 (0.5) | 1.6 (1.3)
  Cass adrenergic score - day 56 (n=5, 6) | 0.6 (0.4) | 1.2 (0.6)

6. Secondary Outcome: Serum Creatinine
Time Frame: baseline, Day 4, Day 7, Day 56
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Hemin | Albumin
Number analyzed (Participants) | 11 | 9
mg/dL
  Baseline | 1.0 (0.1) | 0.7 (0.1)
  Day 4 | 1.0 (0.1) | 0.6 (0.1)
  Day 7 | 0.9 (0.1) | 0.7 (0.1)
  Day 56 | 0.8 (0.1) | 0.7 (0.1)

7. Secondary Outcome: Prothrombin Time
Time Frame: baseline, Day 4, Day 7, Day 56
Measure: Mean (Standard Error); unit: International Normalized Ratio (INR)
Arm/Group | Hemin | Albumin
Number analyzed (Participants) | 11 | 9
International Normalized Ratio (INR)
  Baseline | 1.0 (0.1) | 0.9 (0.1)
  Day 4 | 1.0 (0.1) | 1.0 (0.1)
  Day 7 | 1.0 (0.1) | 1.0 (0.1)
  Day 56 | 1.0 (0.1) | 1.0 (0.1)

8. Secondary Outcome: Activated Partial Thromboplastin Time (APTT)
Time Frame: baseline, Day 4, Day 7, Day 56
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | Hemin | Albumin
Number analyzed (Participants) | 11 | 9
Seconds
  Baseline | 32 (1.8) | 32 (0.9)
  Day 4 | 33 (1.0) | 31 (1.5)
  Day 7 | 30 (1.3) | 31 (1.4)
  Day 56 | 30 (1.2) | 32 (1.3)

9. Secondary Outcome: Hemoglobin
Description: Measured by complete blood count
Time Frame: baseline, Day 4, Day 7, Day 56
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Hemin | Albumin
Number analyzed (Participants) | 11 | 9
g/dL
  Baseline | 12.1 (0.4) | 12.4 (0.5)
  Day 4 | 11.5 (0.5) | 11.5 (0.5)
  Day 7 | 11.6 (0.6) | 11.2 (0.4)
  Day 56 | 11.3 (0.6) | 11.2 (0.3)
Statistical Analysis 1: Comparison: Hemin vs Albumin; Comparison for Day 7; Test type: Superiority or Other; p < 0.05, ANCOVA

10. Secondary Outcome: Erythrocyte Count
Description: Measured by complete blood count
Time Frame: baseline, Day 4, Day 7, Day 56
Measure: Mean (Standard Error); unit: number x 10^12 erythrocytes/L
Arm/Group | Hemin | Albumin
Number analyzed (Participants) | 11 | 9
number x 10^12 erythrocytes/L
  Baseline | 4.1 (0.1) | 4.4 (0.1)
  Day 4 | 4.0 (0.1) | 4.1 (0.1)
  Day 7 | 4.0 (0.2) | 4.0 (0.1)
  Day 56 | 4.0 (0.2) | 4.0 (0.1)
Statistical Analysis 1: Comparison: Hemin vs Albumin; Comparison for Day 7; Test type: Superiority or Other; p < 0.05, ANCOVA

11. Secondary Outcome: Leukocyte and Platelet Counts
Description: Measured by complete blood count
Time Frame: baseline, Day 4, Day 7, Day 56
Measure: Mean (Standard Error); unit: number x 10^9 cells/L
Arm/Group | Hemin | Albumin
Number analyzed (Participants) | 11 | 9
number x 10^9 cells/L
  Leukocytes Baseline | 7.0 (0.6) | 6.0 (0.5)
  Leukocytes Day 4 | 7.0 (0.5) | 6.2 (0.6)
  Leukocytes Day 7 | 7.2 (0.6) | 6.8 (1.2)
  Leukocytes Day 56 | 7.3 (0.5) | 6.5 (0.8)
  Platelets Baseline | 248 (18) | 266 (26)
  Platelets Day 4 | 194 (14) | 246 (21)
  Platelets Day 7 | 201 (15) | 248 (26)
  Platelets Day 56 | 212 (12) | 251 (41)
Statistical Analysis 1: Comparison: Hemin vs Albumin; Comparison for Platelets on Day 4; Test type: Superiority or Other; p = 0.01, ANCOVA

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Hemin | Albumin
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 5/11 | 7/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hemin (N=11) | Albumin (N=9)
Headache (General disorders) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) — Mild to moderate
Dizziness or light headedness (General disorders) | 2 (2) | 0 (0)
Maculopapular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Rash was on both upper extremities

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes